CLINICAL TRIAL: NCT02445716
Title: Transdermal Testosterone Nanoemulsion Effects Emergent Loss of Libido in Women: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Transdermal Testosterone Nanoemulsion in Women Libido
Acronym: Biolipid/B2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Potiguar (Other)
Collaborators: Farmacias Evidence Ltda (Unknown); Lemos laboratório de Análises Clínicas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNIFESP/Evidence
Record Dates: First submitted 2015-05-07; First posted 2015-05-15 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Menopause
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone 500 mcg / Biolipid B2 (Active Comparator): The arm, is part of a randomized, double-blind, placebo-controlled, parallel group trial.
  The arm have 35 women. It consists of a 12-week treatment phase involving three study visits and one telephone contact at week 7 of the treatment.
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): The arm, is part of a randomized, double-blind, placebo-controlled, parallel group trial.
  The arm have 35 women. It consists of a 4-week screening period plus a 12-week treatment phase involving three study visits and one telephone contact at week 7 of the treatment.
  Participants will be attended at the Federal University of São Paulo / Post Graduation Program in São Paulo, Brazil for their study visits.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — It consists of a 12-week treatment with 300mcg of transdermal testosterone phase involving three study visits. Participants will attend at the Federal University of Sao Paulo in Brazil for their study visits.
  Participants will be submitted to a physical examination including vital signs and breast and pelvic examination. Women who met the eligibility criteria is invited to attend a baseline randomization visit. They will be randomly assigned in a 1:1 ratio to receive a transdermal testosterone nanoemulsion (0.8g per dose) delivering 300 mcg/day testosterone or an identical placebo provided by Evidence Pharmaceuticals LTDA, SP, BRAZIL.
  Women are asked to return all unused pumps, and treatment compliance was checked by counting weighting returned packs at their final visit.
  Other Names: Transdermal Testosterone Nanoemulsion
  Arms: Testosterone 500 mcg / Biolipid B2
Drug: Placebo — It consists of a 12-week treatment with placebo phase involving three study visits. Participants will attend at the Federal University of Sao Paulo in Brazil for their study visits.
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled study. Seventy women, aged 35-75 years, with treatment-emergent loss of libido will be randomly allocated to the treatment with a Transdermal nanoemulsion of Testosterone (500mcg) delivering 300 mcg of testosterone/day or an identical placebo nanoemulsion (PLA) for 12 weeks.

DETAILED DESCRIPTION:
The aim of this study is to investigate the efficacy of transdermal testosterone nanoemulsion (TNT) as a treatment for SSRI/SNRI-emergent loss of libido.

The primary outcome measures to be evaluated is the change in the Sabbatsberg Sexual Self-rating Scale (SSS) total score over 12 weeks. The 4-week frequency of Satisfactory Sexual Events (SSEs) and the Female Sexual Distress Scale-Revised (FSDS-R) will be also evaluate.

ELIGIBILITY:
Inclusion Criteria:

* a body mass index between 18 and 27 kg/m2;
* Diminished libido;
* Sexual behavior complaints;
* No evidence of severe clinical depression;
* General good health based on history and physical examination.

Exclusion Criteria:

* a past history of neurological disorder;
* Poor feelings for their partner;
* Had received pharmacotherapy for depression within 8 weeks before screening
* Taking medication known to interfere with normal sexual function (such as α-blockers and β-blockers);
* Recent psychiatric or systemic illness;
* Uncontrolled hypertension (blood pressure>160/95mmHg),
* Unstable cardiovascular disease,
* Genital bleeding;
* Use of psychoactive medications, alcohol excess consumption or any other drug abuse;
* Women who had under gone treatment for acne, depression, dyspareunia.

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Change in sexual function measured by the Sexual Self-rating Scale (SSS) | Baseline and 12 weeks
  The SSS is a 21-item, multiple-choice questionnaire containing seven domains (sexual interest, sexual activity, satisfaction with sexual life, experience of sexual pleasure, sexual fantasy, orgasmic capacity, and sexual relevancy). Each item has five levels scored from 0 to 4. Possible composite scores range from 0 (low sexuality) to 84 (high sexuality). It was developed to use in premenopausal and postmenopausal women .
  Its validity and reliability have been independently established.

CONTACTS AND LOCATIONS:
Overall Officials: Ivaldo Silva, PhD, Study Director — Federal University of São Paulo
Locations (3):
- Brazil (3):
  - Gynelogical Center, Fortaleza, Ceará
  - University Potiguar, Natal, Rio Grande do Norte
  - Marco Botelho, São Paulo

REFERENCES:
- [Result] Botelho MA, Queiroz DB, Barros G, Guerreiro S, Fechine P, Umbelino S, Lyra A, Borges B, Freitas A, Queiroz DC, Ruela R, Almeida JG, Quintans L Jr. Nanostructured transdermal hormone replacement therapy for relieving menopausal symptoms: a confocal Raman spectroscopy study. Clinics (Sao Paulo). 2014 Feb;69(2):75-82. doi: 10.6061/clinics/2014(02)01. PMID 24519196